CLINICAL TRIAL: NCT04682054
Title: Molecular Taxonomy of Surgically-harvested Ocular Tissues Defined by Single-cell Transcriptomics
Acronym: Eyesinglecell
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Eyesinglecell
Record Dates: First submitted 2020-12-07; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Diabetic Retinopathy; Proliferative Vitreoretinopathy; Pterygium; Glaucoma
MeSH Terms: conditions — Diabetic Retinopathy; Vitreoretinopathy, Proliferative; Pterygium; Glaucoma | interventions — Ophthalmologic Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- surgically-removed eye tissue (Experimental)
  Interventions: Procedure: ocular surgery

INTERVENTIONS:
Procedure: ocular surgery — surgery to remove the pathological eye tissue

SUMMARY:
The surgically-harvested eye tissue (ie. vitreous-retinal proliferative membrane, outflow pathway, retinas, and pterygium) is a complex tissue responsible for maintaining intraocular homeostasis or mediating ocular pathogenesis. Dysfunction of one or more resident cell types within the tissues results in different ocular disorder, leading to vision loss, or even blindness. In this study, we aim to use single-cell RNA sequencing to generate a comprehensive cell atlas of surgically-harvested eye tissues.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ocular diseases and require surgery intervention.
2. The surgery intervention remove pathological tissue during surgery.
3. Patients consent to the treatment and single-cell sequencing.

Exclusion Criteria:

1. Surgically removed eye tissue cannot meet with the quality control of single-cell sequencing (mainly the tissue weight and cell counts);

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
counts of each cell type | 1 month
  single-cell sequencing identify what cells and the counts within the eye tissue

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
The single-cell alts of IPD will be available with reasonable request.
Supporting Information: CSR, Analytic Code

REFERENCES:
- [Background] Tan WJ, Wang MM, Castagnoli PR, Tang T, Chan ASY, Lim TS. Single B-Cell Genomic Analyses Differentiate Vitreoretinal Lymphoma from Chronic Inflammation. Ophthalmology. 2021 Jul;128(7):1079-1090. doi: 10.1016/j.ophtha.2020.11.018. Epub 2020 Nov 20. PMID 33221324
- [Background] Wynne N, Carroll J, Duncan JL. Promises and pitfalls of evaluating photoreceptor-based retinal disease with adaptive optics scanning light ophthalmoscopy (AOSLO). Prog Retin Eye Res. 2021 Jul;83:100920. doi: 10.1016/j.preteyeres.2020.100920. Epub 2020 Nov 6. PMID 33161127
- [Background] de Bruijn SE, Fiorentino A, Ottaviani D, Fanucchi S, Melo US, Corral-Serrano JC, Mulders T, Georgiou M, Rivolta C, Pontikos N, Arno G, Roberts L, Greenberg J, Albert S, Gilissen C, Aben M, Rebello G, Mead S, Raymond FL, Corominas J, Smith CEL, Kremer H, Downes S, Black GC, Webster AR, Inglehearn CF, van den Born LI, Koenekoop RK, Michaelides M, Ramesar RS, Hoyng CB, Mundlos S, Mhlanga MM, Cremers FPM, Cheetham ME, Roosing S, Hardcastle AJ. Structural Variants Create New Topological-Associated Domains and Ectopic Retinal Enhancer-Gene Contact in Dominant Retinitis Pigmentosa. Am J Hum Genet. 2020 Nov 5;107(5):802-814. doi: 10.1016/j.ajhg.2020.09.002. Epub 2020 Oct 5. PMID 33022222
- [Background] van Zyl T, Yan W, McAdams A, Peng YR, Shekhar K, Regev A, Juric D, Sanes JR. Cell atlas of aqueous humor outflow pathways in eyes of humans and four model species provides insight into glaucoma pathogenesis. Proc Natl Acad Sci U S A. 2020 May 12;117(19):10339-10349. doi: 10.1073/pnas.2001250117. Epub 2020 Apr 27. PMID 32341164